CLINICAL TRIAL: NCT06173115
Title: The Utilization of Single Versus Double Perclose Devices for Transfemoral Aortic Valve Replacement Access Site Closure: A Prospective, Multicenter, Randomized Controlled Trial
Brief Title: Comparison of a Single Versus Double Perclose Technique for TAVR
Acronym: Single
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAHZJU CT022
Record Dates: First submitted 2023-10-30; First posted 2023-12-15 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Severe Aortic Stenosis
Keywords: transcatheter aortic valve replacement; vascular closure devices; randomized control trial
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Double Perclose device (Active Comparator): Double Perclose device ( Perclose Proglide system, Abbott Vascular) was used for large bore arteriotomy site closure during TF-TAVR procedures
  Interventions: Device: Perclose Proglide system
- Single Perclose device (Experimental): Single Perclose device ( Perclose Proglide system, Abbott Vascular) was used for large bore arteriotomy site closure during TF-TAVR procedures
  Interventions: Device: Perclose Proglide system

INTERVENTIONS:
Device: Perclose Proglide system — "Preclosure" technique has emerged as a common vascular closure approach using a Perclose Proglide system (Abbott Vascular), in which sutures are deployed before dilating the arterial access site.

SUMMARY:
Transcatheter aortic valve replacement (TAVR) has become widely recognized as a minimally invasive approach for aortic valve replacement in patients with severe aortic stenosis. It has been proven to be a safe and effective option for patients who are at low, intermediate, and prohibitive risk for surgical valve replacement.

One of the critical components of procedural success in a transfemoral approach is access site management, as vascular complications strongly correlate with adverse outcomes. When major vascular complications occur, there are higher rates of major bleeding, transfusions, and renal failure requiring dialysis, as well as a significantly higher rate of 30-day and 1-year mortality. In recent years, a "preclosure" technique has emerged as a common vascular closure approach using a Perclose Proglide system (Abbott Vascular), in which sutures are deployed before dilating the arterial access site. This allows for arterial closure after dilation to sizing up to larger bore access sheaths that accommodate valve delivery systems. The sutures are subsequently harvested and tightened to close the large bore arteriotomy site at the end of the case. It has been demonstrated that the use of two Perclose devices, or double Perclose closure, is an effective closure technique with a low rate of vascular complications. A large number of TAVR centers have adopted this method for large-bore vascular closure. In the past, there have been few investigations comparing the utilization of a single Perclose device compared to a double Perclose technique. There are numerous theoretical advantages to the use of a single device, which include decreased procedural cost and procedural time. The investigation aimed to determine if there are clinical benefits as well using the single Perclose approach.

DETAILED DESCRIPTION:
SINGLE-CLOSURE (The utilization of Single versus double perclose devices for transfemoral aortIc valve replacement access site Closure) is an investigator-initiated, open-label, multicenter, randomized controlled trial. The study was approved by the local ethics committees of all participating centers, and each patient provided written informed consent for inclusion in the trial. Data management and analysis was performed by an independent data coordinating center, with oversight from a steering committee. The members of the steering committee had full access to the data and vouch for the accuracy and complete- ness of the data and the analyses. The data that support the findings of this study are available from the corresponding author on reasonable request. Patients scheduled to undergo transfemoral TAVR were considered for inclusion in the trial if they met all inclusion and none of the exclusion criteria. Inclusion criteria were an indication for TAVR as judged by the local heart team; selection of the transfemoral access route and a commercially available transcatheter aortic valve; and willingness to comply with protocol specified follow-up evaluations. Principal exclusion criteria were a vascular access site anatomy not suitable for percutaneous vascular closure and the occurrence of vascular access site complications before the TAVR procedure. Additional exclusion criteria were a known allergy or hypersensitivity to any VCD component; unstable active bleeding or bleeding diathesis or significant unman-ageable anemia; absence of computed tomographic data of the access site before the procedure; systemic infection or a local infection at or near the access site; life expectancy of <6 months because of noncardiac conditions; patients who cannot adhere to or complete the investigational protocol for any reason; pregnant or nursing patients; and participation in any other interventional trial.

The primary end point of the trial was the rate of access site or access-related major and minor vascular complications defined according to the Valve Academic Research Consortium-3 criteria. The end point was assessed during index hospitalization. Relationship to the access site was deter- mined according to the site used for the large-bore vascular access sheath.

Secondary end points included the rate of the primary end point at 30 days; components of the primary end point in-hospital and at 30 days; in-hospital and 30-day major and minor vascular complications; unplanned vascular surgery or use of endovascular stent or stent-graft or other endovascular interventions at the puncture site; in-hospital and 30-day access site- or access-related minor, major, and disabling or life threatening bleeding; need for blood transfusion for access site- or access-related bleeding or vascular complications; rate of VCD failure, defined as the failure of a closure device strategy to achieve hemostasis with the need for an alternative treatment (other than manual compression or adjunctive endovascular ballooning); in-hospital and 30-day all-cause death; in-hospital and 30-day death attributed to access site or access-related complications; need and number of additional unplanned VCDs; time to hemostasis, defined as the time from VCD application to complete hemostasis; and the length of postprocedural hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo transfemoral TAVR were considered for inclusion in the trial if they met all inclusion and none of the exclusion criteria. Inclusion criteria were an indication for TAVR as judged by the local heart team; selection of the transfemoral access route and a commercially available transcatheter aortic valve; and willingness to comply with protocol specified follow-up evaluations.

Exclusion Criteria:

* Principal exclusion criteria were a vascular access site anatomy not suitable for percutaneous vascular closure and the occurrence of vascular access site complications before the TAVR procedure. Additional exclusion criteria were a known allergy or hypersensitivity to any VCD component; unstable active bleeding or bleeding diathesis or significant unman ageable anemia; absence of computed tomographic data of the access site before the procedure; systemic infection or a local infection at or near the access site; life expectancy of <6 months because of noncardiac conditions; patients who can-not adhere to or complete the investigational protocol for any reason; pregnant or nursing patients; and participation in any other interventional trial.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 876 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-28 (Estimated)

PRIMARY OUTCOMES:
The primary end point of the trial was the rate of access site or access-related major and minor vascular complications defined according to the Valve Academic Research Consortium-3 criteria | The end point was assessed during index hospitalization
  1. Aortic dissection or aortic rupture
  2. Vascular (arterial or venous) injury (perforation, rupture, dissection, stenosis, ischaemia, arterial or venous thrombosis including pulmonary embolism, arteriovenous fistula, pseudoaneurysm, haematoma, retroperitoneal haematoma, infection) or compartment syndrome resulting in death, VARC type >_2 bleeding, limb or visceral ischaemia, or irreversible neurologic impairment;
  3. Distal embolization (non-cerebral) from a vascular source resulting in death, amputation, limb or visceral ischaemia, or irreversible endorgan damage;
  4. Unplanned endovascular or surgical intervention resulting in death, VARC type >_2 bleeding, limb or visceral ischaemia, or irreversible neurologic impairment;
  5. Closure device failure c resulting in death, VARC type >_2 bleeding, limb or visceral ischaemia, or irreversible neurologic impairment

SECONDARY OUTCOMES:
The rate of the primary end point at 30 days | 30 days
  the rate of access site or access-related major and minor vascular complications at 30 days
Components of the primary end point in-hospital and at 30 days | 30 days
  Components of the rate of access site or access-related major and minor vascular complications at 30 days
In-hospital and 30-day major and minor vascular complications | 30 days
  In-hospital and 30-day major and minor vascular complications
Unplanned vascular surgery or use of endovascular stent or stent-graft or other endovascular interventions at the puncture site | 30 days
  Unplanned vascular surgery or use of endovascular stent or stent-graft or other endovascular interventions at the puncture site at 30 days
in-hospital and 30-day access site- or access-related minor, major, and disabling or life- threatening bleeding; need for blood transfusion for access site or access related bleeding or vascular complications | 30 days
  in-hospital and 30-day access site- or access-related minor, major, and disabling or life- threatening bleeding; need for blood transfusion for access site or access related bleeding or vascular complications
Rate of VCD failure, defined as the failure of a closure device strategy to achieve hemostasis with the need for an alternative treatment (other than manual compression or adjunctive endovascular ballooning) | 30 days
  Rate of VCD failure, defined as the failure of a closure device strategy to achieve hemostasis with the need for an alternative treatment (other than manual compression or adjunctive endovascular ballooning) at 30 days
In-hospital and 30-day all-cause death; in-hospital and 30-day death attributed to access site- access-related complications; need and number of additional unplanned VCDs | 30 days
  In-hospital and 30-day all-cause death; in-hospital and 30-day death attributed to access site- access-related complications; need and number of additional unplanned VCDs
Time to hemostasis, defined as the time from VCD application to complete hemostasis | 30 days
  Time to hemostasis, defined as the time from VCD application to complete at 30 days
The length of postprocedural hospital stay | 30 days
  The length of postprocedural hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Jianan Wang, PhD, Study Chair — Department of Cardiology, The Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (25):
- China (25):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong
  - Yulin First People's Hospital, Yulin, Guangxi
  - Xiangya Hospital of Central South University, Changshacun, Henan
  - Fuwai Central China Cardiovascular Hospital, Zhengzhou, Henan
  - Henan Provincial Chest Hospital, Zhengzhou, Henan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - General Hospital of Northern Theater Command, PLA, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Qingdao Municipal Hospital, Qingdao, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang
  - Department of Cardiology, The Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Huzhou Central Hospital, Huzhou, Zhejiang
  - Ningbo Medical Center Li Huili Hospital, Ningbo, Zhejiang
  - The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Beijing Anzhen Hospital, Capital Medical University, Beijing
  - Fuwai Hospital, Chinese Academy of Medical Sciences, Beijing

IPD SHARING:
Plan to Share IPD: No